CLINICAL TRIAL: NCT05341388
Title: The Effect of SGLT2 Inhibitors on Cognitive Functions and a Neuroinflammatory Biomarker, Brain-Derived Neurotrophic Factor Levels in Patients With Type 2 Diabetes
Brief Title: The Effect of SGLT2 Inhibitors on Cognitive Functions and BDNF Levels in Patients With Type 2 Diabetes
Status: Terminated | Type: Observational
Why Stopped: not enough participants due to the pandemia
Sponsor: Goztepe Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ayse N Erbakan, MD, Goztepe Training and Research Hospital
Other Study IDs: Cognitive-BDNF
Record Dates: First submitted 2021-10-17; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Type2 Diabetes; Cognitive Impairment
Keywords: type 2 diabetes; cognitive impairment; BDNF; SGLT2 inhibitors
MeSH Terms: conditions — Cognitive Dysfunction; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (2):
- Patients with type 2 diabetes-SGLT2 inh: patients with type 2 diabetes who were recently prescribed an SGLT2 inhibitor
  Interventions: Diagnostic Test: MOCA cognitive evaluation test; Diagnostic Test: BDNF levels; Other: SF-36 test; Diagnostic Test: Geriatric depression test
- Patients with type 2 diabetes-control: patients with type 2 diabetes who were recently prescribed a pre-defined antidiabetic medication other than SGLT2 inhibitors
  Interventions: Diagnostic Test: MOCA cognitive evaluation test; Diagnostic Test: BDNF levels; Other: SF-36 test; Diagnostic Test: Geriatric depression test

INTERVENTIONS:
Diagnostic Test: MOCA cognitive evaluation test — Before starting their newly prescribed medication, we will apply MOCA and repeat it at the end of the trial.
Diagnostic Test: BDNF levels — Before starting their newly prescribed medication, we will apply MOCA and repeat it at the end of the trial.
Other: SF-36 test — Before starting their newly prescribed medication, we will apply MOCA and repeat it at the end of the trial.
Diagnostic Test: Geriatric depression test — Before starting their newly prescribed medication, we will apply MOCA and repeat it at the end of the trial.

SUMMARY:
Cognitive impairment is a common complication in diabetes for various reasons. Although glycemic control improves cognitive impairment, different antidiabetic medications' effects on cognitive functions are still being investigated. Brain-derived neurotrophic factor (BDNF) is a neuroinflammatory marker and a member of the neurotrophin family with growth factor properties. BDNF levels have been shown to decrease in mild cognitive dysfunction or in late-onset Alzheimer's disease. Our aim is to examine the effect of SGLT2 inhibitor use on cognitive functions and BDNF levels.

DETAILED DESCRIPTION:
Type 2 diabetes is a complex metabolic disorder that can cause serious damage to various organs. Impairment in cognitive functions is one of the common complications in patients with diabetes. Impairment in cognitive functions and significant dementia were found to be approximately 1.5 times more common in individuals with diabetes than individuals without diabetes. In particular, inadequate glycemic control, the frequency of hypoglycemia, vascular diseases, insulin resistance, inflammatory cytokines and oxidative stress stand out as possible causes. Brain-derived neurotrophic factor (BDNF) is a member of the neurotrophin family with growth factor properties. BDNF plays a critical role in cell differentiation, migration, and survivable synaptic plasticity of neurons. BDNF also has an important role in learning and memory processes through synapses in the hippocampus. BDNF levels have been shown to decrease in mild cognitive dysfunction or in late-onset Alzheimer's disease. In animal experiments, it has been observed that BDNF values increase with the use of metformin in Parkinson's disease. Similar results were obtained with vildagliptin, alogliptin, rosiglitazone, and exendin-4 in animal experiments.

The effects of drugs used in the treatment of diabetes on protecting or improving cognitive functions have been studied for a long time. Most of these studies are at the preclinical level. In previous studies with Glucagon-Like Peptide 1 (GLP-1) agonists and dipeptidyl peptidase 4 (DPP-4) inhibitors, there are data that both glycemia and incretins improve cognitive functions with their effects on brain structure. Similar positive results are seen for thiazolidinediones. While hyperglycemia control leads to positive results in insulin and sulfonylurea group drugs, the frequency of hypoglycemia can have a negative effect. There is not enough data on SGLT2 inhibitors.

Studies with SGLT2 inhibitors have shown a decrease in HbA1c values, weight loss, and a decrease in both systolic and diastolic blood pressure. Encouraging results have been obtained with SGLT2 inhibitors in both cardiac and renal outcomes, with heart failure in the foreground. As a result of these data, they are recommended as drugs that should be used in the foreground following metformin, especially in diabetic patients with cardiac and renal diseases. Animal studies with empagliflozin and canagliflozin show that both agents reduce cognitive impairment.

Our aim is to examine the effect of SGLT2 inhibitor use on cognitive functions and BDNF, one of the neuroinflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* giving consent
* being 60 years old or older
* HbA1c concentrations between 6.5% and 8%
* using metformin as a single agent for at least 3 months
* diabetes age <10 years

Exclusion Criteria:

* having uncontrolled hypothyroidism, hyperthyroidism, or other diseases that may affect cognitive functions
* ketoacidosis or coma
* cerebrovascular disease or psychiatric disorder
* mental retardation, psychosis, dementia, brain trauma, epilepsy and other cerebral diseases
* alcohol or other substance abuse
* hearing loss
* Presence of diseases that will affect cognitive function such as chronic inflammatory diseases and respiratory system diseases
* chronic kidney failure (GFR <45)
* sleep apnea syndrome
* malignancy
* using a sulfonylurea or glinide

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who refer to a diabetes outpatients clinics to an university hospital
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Cognitive functions | Six months
  We will observe the effects of SGLT2 inhibitors and other oral antidiabetic agents on cognitive functions in type 2 diabetic patients using Montreal Cognitive Assessment (MOCA) test
BDNF concentrations | Six months
  We will observe the effects of SGLT2 inhibitors and other oral antidiabetic agents on BDNF levels in type 2 diabetic patients. We will also assess whether there is an association between cognitive functions and BDNF concentrations in these prespecified groups of patients.

SECONDARY OUTCOMES:
36 item Short Form Survey (SF-36) | Six months
  We will observe the effects of SGLT2 inhibitors and other oral antidiabetic agents on quality of life of life in type 2 diabetic patients using SF-36 survey.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse N Erbakan, MD, Principal Investigator — Istanbul Medeniyet University Goztepe Research and TRaining Hospital; Mehmet Sargın, Prof, Study Chair — Istanbul Medeniyet University; Nazmiye Özbilgin, Prof, Study Chair — University of Health Sciences Siyami Ersek TCS Training and Research Hospital; Aytekin Oğuz, Prof, Study Chair — Istanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University Goztepe Research and Training Hospital, Istanbul, Turkey (Türkiye)